CLINICAL TRIAL: NCT02752646
Title: Tolerability and Toxicity of Topically Applied Nepafenac 0.3% vs Ketorolac 0.5%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDbackline, LLC (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALC-15417759
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Cataract
Keywords: cataract
MeSH Terms: conditions — Cataract | interventions — nepafenac; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nepafenac 0.3% (Active Comparator): Patients in this arm will receive nepafenac 0.3% eye drops once daily following cataract surgery, combined with a topical antibiotic and steroid. This regimen is FDA approved and withing the standard of care.
  Interventions: Drug: nepafenac 0.3%
- ketorolac 0.5% (Active Comparator): Patients in this arm will receive ketorolac 0.5% eye drops four times daily following cataract surgery, combined with a topical antibiotic and steroid. This regimen is FDA approved and withing the standard of care.
  Interventions: Drug: ketorolac

INTERVENTIONS:
Drug: nepafenac 0.3% — Patients in this group will receive nepafenac 0.3% eye drops once daily after cataract surgery.
  Other Names: Ilevro
  Arms: nepafenac 0.3%
Drug: ketorolac — Patients in this group will receive ketorolac 0.5% eye drops four times daily after cataract surgery.
  Arms: ketorolac 0.5%

SUMMARY:
This study will examine the tolerability and toxicity of topically applied Nepafenac 0.3% vs ketorolac 0.5% among patients undergoing cataract surgery.

DETAILED DESCRIPTION:
This will be a randomized, prospective, controlled, open-label study, comparing the tolerability and toxicity of two commercially available non-steroidal anti-inflammatory eye drops, nepafenac 0.3% and ketorolac 0.5% (generic formulation). The study will involve one eye of each subject. The study will follow good clinical practices (GCP). The primary outcome measure will be tolerability of the study medication as measured by the eye drop comfort survey instrument.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years and older currently undergoing femtosecond or manual cataract surgery with or without astigmatic keratotomy.
2. Patients willing to take an electronic survey about their tolerability of either study medication.

Exclusion Criteria

1. Active, systemic or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the questions in the survey and examination findings.
2. Any of the following ocular (eye or eyelid) conditions in either eye within 1 Months prior to the enrollment visit:

   1. Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgery procedure.
   2. Clinically significant ocular trauma.
   3. Active ocular Herpes simplex or Herpes zoster (eye or eyelid) infection.
   4. Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis)
   5. Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye)
3. Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis
4. Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
5. Eyelid abnormalities that significantly affect lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis)
6. Ocular surface abnormality that may compromise corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy)
7. Participation in another ophthalmic clinical trial involving a therapeutic drug or device within 30 days prior to the distribution of the survey
8. Participation in this trial in the same patient's fellow eye.
9. Patients who are pregnant or breastfeeding or who may become pregnant during participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of nepafenac vs ketorolac | 14-28 days
  Patients will fill out a survey describing eye drop tolerability at 14-28 days

CONTACTS AND LOCATIONS:
Overall Officials: John A Hovanesian, MD, Principal Investigator — UCLA Jules Stein Eye Institute
Locations (2):
- United States (2):
  - Harvard Eye Associates, Laguna Hills, California
  - Cincinnati Eye Institute, Edgewood, Kentucky

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual patient data available.

REFERENCES:
- [Result] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Result] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260